CLINICAL TRIAL: NCT05462171
Title: The Prevalence of Erectile Dysfunction (ED) and Premature Ejaculation (PE) in Poland
Acronym: ED POLAND
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Mikolaj Przydacz, Associate Professor, MD PhD DSc PGDip FEBU, Jagiellonian University
Other Study IDs: 1072.6120.331.2021
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Erectile Dysfunction; Premature Ejaculation
MeSH Terms: conditions — Erectile Dysfunction; Premature Ejaculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaires — Participants will be asked to complete validated questionnaires (the five-item International Index of Erectile Function - IIEF-5, Premature Ejaculation Diagnostic Tool - PEDT, International Prostate Symptom Score - IPSS, Overactive Bladder - Validated 8-question Screener - OAB-V8, Hospital Anxiety and Depression Scale - HADS, Athens Insomnia Scale - AIS).

SUMMARY:
The first large population-based study to evaluate erectile dysfunction (ED) and premature ejaculation (PE) in Poland. The study objective is to assess the prevalence and bother of ED and PE in the representative group of male population of Poland.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

• Age <18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A representative group of male Polish population (n=3000).
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of ED in Poland | Through study completion, an average of 3 months
  The prevalence of ED will be assessed using the five-item International Index of Erectile Function (IIEF-5; the lowest score 5; the highest score 25; the lower the score, the greater the severity of the symptoms)
Prevalence of PE in Poland | Through study completion, an average of 3 months
  The prevalence of PE will be assessed using the Premature Ejaculation Diagnostic Tool (PEDT; the lowest score 0; the highest score 20; the lower the score, the lower the severity of the symptoms)

SECONDARY OUTCOMES:
Bother of ED and PE in Poland | Through study completion, an average of 3 months
  The degree of associated bother will be assessed using Likert scale (Likert scale: delighted [score 0], pleased [score 1], mostly satisfied [score 2], mixed [score 3], mostly dissatisfied [score 4], unhappy [score 5], or terrible [score 6]).
Prevalence of lower urinary tract symptoms in patients with PE and ED in Poland | Through study completion, an average of 3 months
  The prevalence of lower urinary tract symptoms will be assessed with the International Prostate Symptom Score (IPSS; the lowest score 0, the highest score 35, the lower the score, the lower the severity of the symptoms)
Prevalence of overactive bladder in patients with PE and ED in Poland | Through study completion, an average of 3 months
  The prevalence of overactive bladder will be assessed with the Overactive Bladder - Validated 8-question Screener (OAB-V8; the lowest score 0; the highest score 40; the lower the score, the lower the severity of the symptoms)
Prevalence of depressive symptoms in patients with PE and ED in Poland | Through study completion, an average of 3 months
  The prevalence of depressive symptoms will be assessed with the Hospital Anxiety and Depression Scale (HADS; the lowest score 0; the highest score 48; the lower the score, the lower the severity of the symptoms)
Prevalence of insomnia in patients with PE and ED in Poland | Through study completion, an average of 3 months
  The prevalence of insomnia will be assessed with the Athens Insomnia Scale (AIS; the lowest score 0; the highest score 24; the lower the score, the lower the severity of the symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

REFERENCES:
- [Derived] Przydacz M, Rajwa P, De Cillis S, Guillot-Tantay C, Herve F, Tienza Fernandez A, Tutolo M, Culha MG, Geretto P, Shenhar C, Miszczyk M, Chlosta P, Phe V, Osman N; European Association of Urology Young Academic Urologists (EAU YAU) Functional Urology Working Group. Lower Urinary Tract Symptoms Correlate with Erectile Dysfunction and Premature Ejaculation but Not with Men's Sexual Activity: Results from a Large Population-Representative Study. Healthcare (Basel). 2024 Jul 15;12(14):1408. doi: 10.3390/healthcare12141408. PMID 39057551